CLINICAL TRIAL: NCT07387419
Title: Ultradian Steroid Rhythms in Adrenal Incidentalomas.
Acronym: CHRONOMACS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2025/067
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Mild Autonomous Cortisol Secretion Adenoma; Non Secreting Adenoma
Keywords: Adrenal incidentaloma; Mild autonomous cortisol secretion adenoma; Ultradian steroid rhythms
MeSH Terms: conditions — Adrenal incidentaloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MACS patients (Experimental): Analysis of the dynamics/rhythmicity of interstitial cortisol and other steroid concentrations thanks to U-RHYTHM system, in MACS patients
  Interventions: Device: U-RYTHM system
- ANS patients (Active Comparator): Analysis of the dynamics/rhythmicity of interstitial cortisol and other steroid concentrations thanks to an original and innovative U-RHYTHM system, interstitial fluid samples, in ANS patients
  Interventions: Device: U-RYTHM system

INTERVENTIONS:
Device: U-RYTHM system — Consent will be obtained at inclusion. The patient will be seen by the investigating physician twice, 27 hours apart, for insertion and removal of the U-RHYTHM system. Microdialysis samples will be collected in the collection system. Samples will be directly frozen at -20°C or -80°C and transported at -20°C to the Ultradian Analysis Laboratory, Metabolomics Centre, Department of Clinical Sciences, University of Bergen, Norway, for sample preparation, LC-MSMS steroid profiling (panel of 21 steroids) and statistical analysis. The research protocol does not include patient follow-up.

SUMMARY:
Twenty to 40% of adrenal incidentalomas are responsible for MACS (mild autonomous cortisol producing secretion). The biological tools used in current practice to explore MACS do not provide precise information on cortisol production abnormalities. This study is a comparative analysis of the dynamics/rhythmicity of interstitial cortisol and other steroid concentrations between MACS and non-secreting adenomas (ANS). Using the original and innovative U-RHYTHM system, interstitial fluid samples will be taken every 20 minutes for 24 to 48 hours from patients with MACS or non-secreting adenomas, and steroid assays will be performed in the perfusates to analyze steroid hormone production over 24 hours.

DETAILED DESCRIPTION:
Adrenal incidentalomas are adrenal masses discovered incidentally during abdominal imaging. They are benign in the vast majority of cases, and most often non-secreting (non-secreting adenoma or ANS). In around 30% of cases, they are responsible for autonomous and moderately excessive cortisol secretion (MACS for "mild autonomous cortisol secretion"). MACS are associated with an increased prevalence of cardiovascular and metabolic comorbidities, and higher mortality than ANS. Beyond the quantitative cortisol production, that serves as a clock for biological rhythm of multiples organs (muscle, liver etc.), the integrity of the cortisol "nadir" (minimal levels around midnight) is fundamental from a metabolic perspective. As cortisol hypersecretion in MACS is moderate, it is suggested that its impact is linked to qualitative/temporal abnormalities in the secretion of cortisol and/or other related steroids. Only two studies (Debono, JCEM, 2017; Ceccato, Endocrine, 2018) suggest that excessive cortisol production in MACS may occur in the late afternoon or early evening. However, these studies are based on a small number of subjects and are hampered by the small number of blood or saliva samples, which are inappropriate to accurately assess the dynamics of daily cortisol secretion. In addition, these studies do not address the dynamics of other adrenal steroids that may play a role in the pathophysiology of MACS. The U-RHYTHMS sampling system is an original and innovative system for analyzing the dynamics of steroid hormone production over 24 hours. Using interstitial fluid samples taken every 20 min for 24 to 48 hours, in which hormone assays are performed, we will study the 24-hour steroid production dynamics in MACS and compare it with that of ANS. Apart from a pathophysiological interest, a better understanding of the abnormal dynamics of cortisol production could improve firstly the diagnostic of MACS with the identification of target periods to perform blood samples ; and, secondly, improve therapeutic management of patients with the identification of appropriate periods for the administration of short-acting steroidogenic drugs.

Consent will be obtained at inclusion. The patient will be seen by the investigating physician twice, 27 hours apart, for insertion and removal of the U-RHYTHM system. Microdialysis samples will be collected in the collection system. Samples will be directly frozen at -20°C or -80°C and transported at -20°C to the Ultradian Analysis Laboratory, Metabolomics Centre, Department of Clinical Sciences, University of Bergen, Norway, for sample preparation, LC-MSMS steroid profiling (panel of 21 steroids) and statistical analysis. The research protocol does not include patient follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18 < Age ≤ 85 years.
* Patient with one or more uni or bilateral adrenal nodules of cortical appearance on CT scan.
* Subject affiliated or beneficiary of a social security scheme.

The diagnostic criteria are:

For the MACS group:

* a serum cortisol concentration after a minute braking test with dexamethasone > 50 nmol/L or 1.8 µg/dL, with a concomitant dexamethasone concentration above the test validation threshold
* morning plasma ACTH concentration ≤ 2.5 pmol/L or 11 pg/mL.

For the non-secreting adenoma group:

- Plasma cortisol after minute dexamethasone braking test ≤ 50 nmol/L or 1.8 µg/dL.

Exclusion Criteria:

* Age < 18 years
* Pregnant or breast-feeding
* Use of oral estrogens (must be discontinued for at least 6 weeks prior to sampling)
* Known adrenal insufficiency and/or treatment with steroids (oral, inhaled, parenteral or topical) or other interfering drugs.
* patient taking part in another study
* Patients placed under legal protection measures and/or deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Rhythm and intensity of cortisol production | During day 1
  The primary outcome is a composite endpoint based on the calculation of five numerical biomarkers of cortisol:
  (i) area under the curve (AUC) during the day (6:00-18:00) ; (ii) AUC during the night (6:00 p.m. to 6:00 a.m.); (iii) peak-to-nadir ratio (PNR) between morning peak (3:00-12:00) and night nadir; (iv) night nadir time (NNT); (v) morning peak time (MPT).

SECONDARY OUTCOMES:
Assessment of the rhythm and intensity of cortisone production | During day 1
  The secondary outcome is a composite endpoint based on the calculation of five numerical biomarkers of cortisone:
  (i) area under the curve (AUC) during the day (6:00-18:00) ; (ii) AUC during the night (6:00 p.m. to 6:00 a.m.); (iii) peak-to-nadir ratio (PNR) between morning peak (3:00-12:00) and night nadir; (iv) night nadir time (NNT); (v) morning peak time (MPT).
Assessment of the rhythm and intensity of 18hydroxycortisol production | During day 1
  The secondary outcome is a composite endpoint based on the calculation of five numerical biomarkers of 18hydroxycortisol:
  (i) area under the curve (AUC) during the day (6:00-18:00) ; (ii) AUC during the night (6:00 p.m. to 6:00 a.m.); (iii) peak-to-nadir ratio (PNR) between morning peak (3:00-12:00) and night nadir; (iv) night nadir time (NNT); (v) morning peak time (MPT).
Assessment of the rhythm and intensity of dehydroandrosténédione production | During day 1
  The secondary outcome is a composite endpoint based on the calculation of five numerical biomarkers of dehydroandrosténédione sulfate (SDHEA):
  (i) area under the curve (AUC) during the day (6:00-18:00) ; (ii) AUC during the night (6:00 p.m. to 6:00 a.m.); (iii) peak-to-nadir ratio (PNR) between morning peak (3:00-12:00) and night nadir; (iv) night nadir time (NNT); (v) morning peak time (MPT).
Assessment of the rhythm and intensity of allo-tetrahydrocortisol production | During day 1
  The secondary outcome is a composite endpoint based on the calculation of five numerical biomarkers of allo-tetrahydrocortisol: (i) area under the curve (AUC) during the day (6:00-18:00) ; (ii) AUC during the night (6:00 p.m. to 6:00 a.m.); (iii) peak-to-nadir ratio (PNR) between morning peak (3:00-12:00) and night nadir; (iv) night nadir time (NNT); (v) morning peak time (MPT).
Assessment of the rhythm and intensity of tetrahydrocortisol production | During day 1
  The secondary outcome is a composite endpoint based on the calculation of five numerical biomarkers of other steroids tetrahydrocortisol (THF):
  (i) area under the curve (AUC) during the day (6:00-18:00) ; (ii) AUC during the night (6:00 p.m. to 6:00 a.m.); (iii) peak-to-nadir ratio (PNR) between morning peak (3:00-12:00) and night nadir; (iv) night nadir time (NNT); (v) morning peak time (MPT).
Assessment of the rhythm and intensity of aldosterone production | During day 1
  The secondary ourcome is a composite endpoint based on the calculation of five numerical biomarkers of other steroids aldosterone:
  (i) area under the curve (AUC) during the day (6:00-18:00) ; (ii) AUC during the night (6:00 p.m. to 6:00 a.m.); (iii) peak-to-nadir ratio (PNR) between morning peak (3:00-12:00) and night nadir; (iv) night nadir time (NNT); (v) morning peak time (MPT).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Haut-Levêque, Pessac, France